CLINICAL TRIAL: NCT03811912
Title: A Randomized Parallel-Group Study to Evaluate the Efficacy and Tolerability of Two Dosing Regimens of CTP-543 in Adult Patients With Moderate to Severe Alopecia Areata
Brief Title: Efficacy and Tolerability Study of Two Dose Regimens of CTP-543 in Adults With Alopecia Areata
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Concert Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CP543.2002
Record Dates: First submitted 2019-01-18; First posted 2019-01-22 (Actual); Results first posted 2022-12-09 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-11

CONDITIONS: Alopecia Areata
MeSH Terms: conditions — Alopecia Areata

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CTP-543 8 mg BID (Experimental): Participants received 1 x 8 mg CTP-543 tablet and 1 x CTP-543 matching placebo tablet, twice daily (BID) for 24 weeks.
  Interventions: Drug: CTP-543; Drug: CTP-543 Matching Placebo
- CTP-543 16 mg QD (Experimental): Participants received 16 mg (2 x 8 mg) CTP-543 tablets, once daily (QD) and after 12 hours, received 2 x CTP-543 matching placebo tablets, QD for 24 weeks.
  Interventions: Drug: CTP-543; Drug: CTP-543 Matching Placebo

INTERVENTIONS:
Drug: CTP-543 — CTP-543 administered as 8 mg tablet.
Drug: CTP-543 Matching Placebo — Administered as tablets to aid treatment masking.

SUMMARY:
This study will evaluate the efficacy and tolerability of once-daily versus twice-daily dosing of CTP-543, in adult patients with chronic, moderate to severe alopecia areata.

ELIGIBILITY:
Inclusion Criteria:

* Definitive diagnosis of alopecia areata with a current episode lasting at least 6 months and not exceeding 10 years at the time of Screening. Total disease duration greater than 10 years is permitted.
* At least 50% scalp hair loss, as defined by a Severity of Alopecia Tool (SALT) score ≥50, at Screening and Baseline.
* Clinical lab results within the normal range

Exclusion Criteria:

* Active scalp inflammation, psoriasis, or seborrheic dermatitis requiring topical treatment to the scalp, significant trauma to the scalp, or untreated actinic keratosis on the scalp.
* Treatment with systemic immunosuppressive medications or biologics.
* Vaccination with herpes zoster vaccine or any live virus within 6 weeks of screening or during the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2019-03-21 (Actual); Primary Completion 2019-11-21 (Actual); Study Completion 2019-11-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Colleen E Hamilton, MS, Study Director — Concert Pharmaceuticals, Inc.
Locations (9):
- United States (9):
  - Investigative Site, Irvine, California
  - Investigative Site, San Francisco, California
  - Investigative Site, New Haven, Connecticut
  - Investigative Site, Boynton Beach, Florida
  - Investigative Site, Boston, Massachusetts
  - Investigative Site, Fridley, Minnesota
  - Investigative Site, Portsmouth, New Hampshire
  - Investigative Site, Winston-Salem, North Carolina
  - Investigative Site, Portland, Oregon

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 10 study centers in the United States from 21 March 2019 to 21 November 2019.
Pre-assignment Details: 70 participants were screened out of which 57 participants who experienced an episode of hair loss due to alopecia areata were enrolled and randomized to receive CTP-543 8 mg twice daily (BID) or CTP-543 16 mg once daily (QD).
Groups:
- CTP-543 8 mg BID: Participants received 1 x 8 mg CTP-543 tablet and 1 x CTP-543 matching placebo tablet, BID for 24 weeks.
- CTP-543 16 mg QD: Participants received 16 mg (2 x 8 mg) CTP-543 tablets, QD and after 12 hours, received 2 x CTP-543 matching placebo tablets, QD for 24 weeks.
Period: Overall Study
Arm/Group | CTP-543 8 mg BID | CTP-543 16 mg QD
Started | 29 | 28
Safety Population (Safety Population included all participants who received study drug. Participants in the safety population were analyzed according to the actual dosing regimen received during the study.) | 29 | 28
Completed | 25 | 26
Not Completed | 4 | 2
Not completed — Withdrew Consent | 4 | 2

BASELINE CHARACTERISTICS:
Population: Randomized Population included all the randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | CTP-543 8 mg BID | CTP-543 16 mg QD | Total
Number analyzed (Participants) | 29 | 28 | 57
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.4 (12.98) | 39.8 (13.65) | 40.1 (13.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 18 | 38
  Male | 9 | 10 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 4 | 7
  Not Hispanic or Latino | 26 | 24 | 50
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 0 | 0 | 0
  Race: Asian | 2 | 1 | 3
  Race: Black or African American | 0 | 3 | 3
  Race: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Race: White | 27 | 23 | 50
  Race: Other | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 29 | 28 | 57
Severity of Alopecia Tool (SALT) Score [Mean (Standard Deviation); unit: score on a scale] — The SALT is a quantitative assessment of scalp hair loss. SALT scores range in severity from 0 (no hair loss) to a maximum of 100 (complete hair loss).
  score on a scale | 87.1 (17.23) | 90.4 (17.46) | 88.7 (17.27)

OUTCOME MEASURES:

1. Primary Outcome: Relative Change From Baseline in Severity of Alopecia Tool (SALT) Score at Week 24
Description: The SALT is a quantitative assessment of scalp hair loss. SALT scores range in severity from 0 (no hair loss) to a maximum of 100 (complete hair loss). Relative change (percent change) to baseline is calculated as: 100 x ([baseline SALT score - follow-up SALT score]/baseline SALT score).
Time Frame: Baseline, Week 24
Population: Efficacy Population included all participants who received study drug and had at least 1 post-treatment SALT assessment. Participants in the efficacy population were analyzed according to their randomized dosing regimen.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | CTP-543 8 mg BID | CTP-543 16 mg QD
Number analyzed (Participants) | 29 | 28
percent change | 46.4 (38.21) | 18.0 (32.32)

2. Secondary Outcome: Percentage of Participants Achieving at Least a 90%, 75%, and 50% Relative Reduction in SALT Score From Baseline
Description: The SALT is a quantitative assessment of scalp hair loss. SALT scores range in severity from 0 (no hair loss) to a maximum of 100 (complete hair loss). Percentage of participants achieving at least a 50%, 75%, 90% relative reduction in SALT score from baseline at Weeks 4, 8, 12, 16, 20, and 24 are reported.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, and 24
Population: as for outcome 1
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | CTP-543 8 mg BID | CTP-543 16 mg QD
Number analyzed (Participants) | 29 | 28
Percentage of participants
  90% Reduction: Week 4 | 0 [0 to 1.7] | 0 [0 to 1.8]
  90% Reduction: Week 8 | 0 [0 to 1.7] | 0 [0 to 1.8]
  90% Reduction: Week 12 | 3.4 [0 to 10.7] | 0 [0 to 1.8]
  90% Reduction: Week 16 | 6.9 [0 to 16.4] | 0 [0 to 1.8]
  90% Reduction: Week 20 | 13.8 [1.5 to 26.0] | 0 [0 to 1.8]
  90% Reduction: Week 24 | 20.7 [6.6 to 34.8] | 3.6 [0 to 11.1]
  75% Reduction: Week 4 | 0 [0 to 1.7] | 0 [0 to 1.8]
  75% Reduction: Week 8 | 3.4 [0 to 10.7] | 3.6 [0 to 11.1]
  75% Reduction: Week 12 | 6.9 [0 to 16.4] | 0 [0 to 1.8]
  75% Reduction: Week 16 | 20.7 [6.6 to 34.8] | 3.6 [0 to 11.1]
  75% Reduction: Week 20 | 31.0 [15.2 to 46.9] | 10.7 [0 to 22.1]
  75% Reduction: Week 24 | 31.0 [15.2 to 46.9] | 10.7 [0 to 22.1]
  50% Reduction: Week 4 | 0 [0 to 1.7] | 0 [0 to 1.8]
  50% Reduction: Week 8 | 6.9 [0 to 16.4] | 3.6 [0 to 11.1]
  50% Reduction: Week 12 | 24.1 [9.3 to 38.9] | 7.1 [0 to 16.9]
  50% Reduction: Week 16 | 34.5 [18.2 to 50.7] | 14.3 [1.6 to 26.9]
  50% Reduction: Week 20 | 41.4 [24.6 to 58.1] | 14.3 [1.6 to 26.9]
  50% Reduction: Week 24 | 48.3 [31.3 to 65.3] | 17.9 [4.2 to 31.5]

3. Secondary Outcome: Absolute Change in SALT Scores From Baseline at Weeks 4, 8, 12, 16, 20, and 24
Description: The SALT is a quantitative assessment of scalp hair loss. SALT scores range in severity from 0 (no hair loss) to a maximum of 100 (complete hair loss). Absolute change equals the difference in SALT measurements (baseline SALT score - follow-up SALT score).
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, and 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | CTP-543 8 mg BID | CTP-543 16 mg QD
Number analyzed (Participants) | 29 | 28
Score on a scale
  Change from Baseline at Week 4 | 0.8 (6.92) | -0.8 (4.49)
  Change from Baseline at Week 8 | 6.5 (15.02) | 2.1 (11.93)
  Change from Baseline at Week 12 | 18.5 (23.27) | 5.3 (19.48)
  Change from Baseline at Week 16 | 27.0 (29.31) | 9.4 (25.46)
  Change from Baseline at Week 20 | 32.8 (29.25) | 13.4 (28.06)
  Change from Baseline at Week 24 | 37.7 (30.75) | 15.7 (28.25)

4. Secondary Outcome: Relative Change in SALT Scores From Baseline at Weeks 4, 8, 12, 16 and 20
Description: as for outcome 1
Time Frame: Baseline, Weeks 4, 8, 12, 16 and 20
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | CTP-543 8 mg BID | CTP-543 16 mg QD
Number analyzed (Participants) | 29 | 28
percent change
  Change from Baseline at Week 4 | 1.4 (9.67) | -1.3 (7.26)
  Change from Baseline at Week 8 | 8.6 (20.58) | 2.7 (19.43)
  Change from Baseline at Week 12 | 23.7 (31.25) | 5.1 (22.91)
  Change from Baseline at Week 16 | 33.3 (35.90) | 9.4 (28.85)
  Change from Baseline at Week 20 | 40.6 (36.85) | 14.8 (31.26)

5. Secondary Outcome: Percentage of Participants With Change in Satisfaction of Hair Coverage
Description: Participant satisfaction question was used to assess overall satisfaction with hair coverage, with responses ranging from 1 to 5, as follows: 1 (very dissatisfied), 2 (dissatisfied), 3 (somewhat satisfied), 4 (mostly satisfied), 5 (very satisfied). Higher scores indicate better satisfaction with hair coverage. The percentage of participants with change from Baseline to the Week 24 satisfaction level was reported as categories: satisfied to satisfied; satisfied to dissatisfied; dissatisfied to satisfied and dissatisfied to dissatisfied. Data is reported only for participants with change from Baseline in satisfaction level.
Time Frame: Baseline, Week 24
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | CTP-543 8 mg BID | CTP-543 16 mg QD
Number analyzed (Participants) | 29 | 28
Percentage of participants
  Satisfied to Satisfied | 0 | 3.6
  Satisfied to Dissatisfied | 3.4 | 0
  Dissatisfied to Satisfied | 55.2 | 17.9
  Dissatisfied to Dissatisfied | 34.5 | 75.0

6. Other Pre Specified Outcome: Number of Participants With Adverse Events as a Measure of Safety
Time Frame: 24 Weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse Events: From first dose of study drug up to Week 28; All-cause mortality: Randomization up to Week 28
Description: Safety Population included all participants who received study drug during the treatment period. Participants were analyzed according to the actual treatment received during the study.
Arm/Group | CTP-543 8 mg BID | CTP-543 16 mg QD
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/28
Other Adverse Events (participants affected / at risk) | 23/29 | 23/28
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CTP-543 8 mg BID (N=29) | CTP-543 16 mg QD (N=28)
Nasopharyngitis (Infections and infestations) | 5 | 5
Upper respiratory tract infection (Infections and infestations) | 5 | 3
Constipation (Gastrointestinal disorders) | 3 | 1
Nausea (Gastrointestinal disorders) | 2 | 0
Acne (Skin and subcutaneous tissue disorders) | 4 | 4
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 2
Fall (Injury, poisoning and procedural complications) | 0 | 2
Headache (Nervous system disorders) | 8 | 5
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Weight increased (Investigations) | 1 | 3
Anxiety (Psychiatric disorders) | 2 | 1
Increased tendency to bruise (Blood and lymphatic system disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an Investigator wants to publish study data or results, the publication or presentation must be provided to Concert for review at least 60 days in advance. If Concert needs to file a patent application prior to publication, the publication can be delayed up to 90 days from Sponsor providing notice to the investigator of such need.

DOCUMENTS (2):
  • Study Protocol (2019-01-03): https://cdn.clinicaltrials.gov/large-docs/12/NCT03811912/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-11): https://cdn.clinicaltrials.gov/large-docs/12/NCT03811912/SAP_001.pdf